CLINICAL TRIAL: NCT01411137
Title: An Open Label Conversion Study of Carbidopa-Levodopa (CD-LD) Extended-Release Taken Alone or in Combination With CD-LD Immediate Release to IPX066 Followed by an Open-Label Extension Safety Study of IPX066 in Advanced PD
Brief Title: Carbidopa-Levodopa (CD-LD) ER Alone or in Combination With CD-LD IR to IPX066 Followed by IPX066 Extension Safety Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPX066-B11-01
Record Dates: First submitted 2011-08-04; First posted 2011-08-08 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2017-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IPX066 (Experimental): Subjects were to receive individualized IPX066 doses orally in an open-label manner using four dosage strengths.
  Interventions: Drug: IPX066

INTERVENTIONS:
Drug: IPX066 — Subjects were converted from their current treatment to IPX066 over a 6-week period.
  Experimental Drug Product: IPX066 (carbidopa-levodopa) extended-release capsules
  Other Names: ER CD-LD

SUMMARY:
The study had three distinct parts and is described as follows:

Part 1:

* To evaluate the dose conversion from CD-LD ER taken alone or in combination with CD-LD IR to IPX066 in subjects with advanced PD
* To evaluate the utility of the Objective Parkinson's Disease Measurement (OPDM), an exploratory computer-based system, in assessing dexterity and mobility in a subset of PD subjects.

Part 2:

• To evaluate the long-term safety and clinical utility of IPX066 under open-label conditions in eligible subjects who successfully completed Part 1 of the study.

Part 3:

• To further evaluate the long-term safety of IPX066 in eligible subjects who successfully completed Part 2.

DETAILED DESCRIPTION:
Part 1: This study was a multicenter, open-label study. Subjects were to be converted from their previous CD-LD treatment to IPX066 over a 6-week period. Up to 40 subjects were to be enrolled in the study. Enrollment was defined as subjects who received study drug in Part 1 - Visit 1. Subjects were to be entered into one of two cohorts.

Approximately 24 subjects were to enroll in Cohort 1 (non-OPDM subjects) and up to 16 subjects at selected sites were to enroll in Cohort 2 (OPDM subjects). For the subjects enrolled in Cohort 2, along with the OPDM measurements, PK blood samples were also to be collected.

Part 2: Following the successful completion of Part 1 of the study, eligible subjects could participate in Part 2, a 6-month open-label extension study.

Part 3: Following the successful completion of Part 2 of the study, eligible subjects could participate in Part 3, an additional 6-month open-label extension study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with idiopathic PD without any known cause for Parkinsonism.
2. At least 30 years old at the time of PD diagnosis.
3. Currently being treated with:

   * an LD dosing frequency of at least four times a day
   * at least one dose of CD-LD ER daily
   * requiring a total daily LD dose of at least 400 mg
   * stable regimen for at least 4 weeks prior to Screening
4. Concomitant therapy with amantadine, anticholinergics, selective monoamine oxidase (MAO) type B inhibitors (e.g., selegiline, rasagiline) or dopamine agonists is allowed as long as the doses and regimens have been stable for at least 4 weeks prior to Screening and the therapy is intended to be constant throughout the course of the study.
5. Agrees to use a medically acceptable method of contraception throughout the study and for 1 month after completing the study.

Exclusion Criteria:

1. Pregnant or breastfeeding
2. Diagnosed with atypical Parkinsonism or any known secondary Parkinsonian syndrome.
3. Nonresponsive to LD therapy.
4. Prior functional neurosurgical treatment for PD (e.g., ablation or deep brain stimulation) or if such procedures are anticipated during study participation.
5. Planning to take during participation in the clinical study: any controlled-release LD product, additional CD or benserazide, entacapone or tolcapone, nonselective MAO inhibitors, or antipsychotics including neuroleptic agents for the purpose of treating psychosis or bipolar disorder.
6. Any evidence of suicidal behavior within 6 months of entering the study.
7. Allergic or hypersensitive to to CD, LD, entacapone, riboflavin, Yellow Dye #5 (tartrazine), citrus fruit or grape juice.
8. History of or currently active psychosis.
9. Active or history of peptic ulcers or surgical procedure of the stomach, the small intestine or the large intestine.
10. Active or history of narrow-angle glaucoma.
11. History of malignant melanoma or a suspicious undiagnosed skin lesion.
12. History of myocardial infarction with residual atrial, nodal, or ventricular arrhythmias, upper gastrointestinal hemorrhage, or neuroleptic malignant syndrome and/or nontraumatic rhabdomyolysis.
13. Abnormal kidney function
14. Severe hepatic impairment.
15. Received any investigational medications during the 4 weeks prior to Screening.
16. Previously enrolled in IPX066 studies.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Impax Study Director, Study Chair — Impax Laboratories, LLC
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Coastal Neurological Medical Group, La Jolla, California
  - The Parkinson's Institute, Sunnyvale, California
  - Renstar Medical Research, Ocala, Florida
  - Quest Research Institute, Bingham Farms, Michigan
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Parkinson's Disease and Movement Disorders Center of Long Island, Commack, New York
  - Wisconsin Institute for Neurologic and Sleep Disorders, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tetrud J, Nausieda P, Kreitzman D, Liang GS, Nieves A, Duker AP, Hauser RA, Farbman ES, Ellenbogen A, Hsu A, Kell S, Khanna S, Rubens R, Gupta S. Conversion to carbidopa and levodopa extended-release (IPX066) followed by its extended use in patients previously taking controlled-release carbidopa-levodopa for advanced Parkinson's disease. J Neurol Sci. 2017 Feb 15;373:116-123. doi: 10.1016/j.jns.2016.11.047. Epub 2016 Nov 23. PMID 28131167

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date first subject enrolled: August 19, 2011 Date last subject completed: March 20, 2013
Groups:
- IPX066: extended-release CD-LD
Period: Part 1: Dose Conversion
Arm/Group | IPX066
Started | 43
Completed | 33
Not Completed | 10
Period: Part 2: Open-Label Extension
Arm/Group | IPX066
Started | 32 (1 subject who completed Part 1 did not elect to continue into Part 2.)
Completed | 25
Not Completed | 7
Period: Part 3: Open-Label Extension
Arm/Group | IPX066
Started | 12 (Two sites with 11 completers of Part 2 did not participate in Part 3. Two subjects lost contact.)
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Subjects converted from their previous CD-LD treatment to IPX066 over a 6-week period.
  Following the successful completion of Part 1 of the study, eligible subjects could participate in Part 2, a 6-month open-label extension study.
  Following the successful completion of Part 2 of the study, eligible subjects could participate in Part 3, an additional 6-month open-label extension study.
Arm/Group | All Study Participants
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Patient Global Impression (PGI)
Description: At Part 1 Week 6, Part 2 Month 3 and Month 6 or at Early Termination, the subjects rated the change in their condition with IPX066 treatment from their condition prior to Part 1 Visit 1(Baseline) using Patient Global Impression (PGI) 7-point scale. 1=very much worse and 7=very much improved.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Part 1: Conversion: Subjects converted from their previous CD-LD treatment to IPX066 over a 6-week period.
- Part 2: Open-Label Extension (Month 3); Part 2: Open-Label Extension (Month 6): Following the successful completion of Part 1 of the study, eligible subjects could participate in Part 2, a 6-month open-label extension study.
- Part 1 or 2 Early Termination: Subjects converted from their previous CD-LD treatment to IPX066 over a 6-week period.
  Following the successful completion of Part 1 of the study, eligible subjects could participate in Part 2, a 6-month open-label extension study.
Arm/Group | Part 1: Conversion | Part 2: Open-Label Extension (Month 3) | Part 2: Open-Label Extension (Month 6) | Part 1 or 2 Early Termination
Number analyzed (Participants) | 33 | 26 | 25 | 15
units on a scale | 5.2 (1.35) | 5.4 (1.30) | 5.3 (1.49) | 2.8 (1.21)

2. Primary Outcome: Clinical Global Impression (CGI)
Description: Clinician-reported satisfaction outcome of IPX066 using Clinical Global Impression (PGI) 7-point scale.
  At Part 1 Week 6; Part 2 Month 3, and Month 6 or at Early Termination, the Investigator rated how much a subject's overall condition had changed since Part 1 Visit 1 (Baseline) using 7-point scale. 1=very much worse and 7=very much improved.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1: Conversion | Part 2: Open-Label Extension (Month 3) | Part 2: Open-Label Extension (Month 6) | Part 1 or 2 Early Termination
Number analyzed (Participants) | 33 | 26 | 25 | 15
units on a scale | 5.5 (1.15) | 5.7 (1.08) | 5.6 (1.39) | 3.7 (0.80)

3. Primary Outcome: Parkinson's Disease Questionnaire-8 (PDQ-8)
Description: Change from Baseline in Parkinson's disease Questionnaire-8 (PDQ-8) at End of Study or early discontinuation. The PDQ-8 is a self-reported questionnaire consisting of 8 questions regarding the subject's disease symptoms, each item ranging from 0 to 4, and the responses consist of 0=Never, 1=Occasionally, 2=Sometimes, 3=Often, and 4=Always or cannot do at all, total score ranging from 0 (never have problems/issues) to 32 (always have problems or cannot do at all).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Part 1: Conversion (Baseline); Part 1: Conversion (Week 6): Subjects converted from their previous CD-LD treatment to IPX066 over a 6-week period.
Arm/Group | Part 1: Conversion (Baseline) | Part 1: Conversion (Week 6) | Part 2: Open-Label Extension (Month 3) | Part 2: Open-Label Extension (Month 6) | Part 1 or 2 Early Termination
Number analyzed (Participants) | 43 | 33 | 26 | 25 | 15
units on a scale | 9.6 (5.49) | 8.1 (4.62) | 8.5 (4.79) | 9.0 (5.91) | 11.8 (6.62)

ADVERSE EVENTS:
Time Frame: 58 weeks
Groups:
- Part 2: Open-Label Extension 1: Following the successful completion of Part 1 of the study, eligible subjects could participate in Part 2, a 6-month open-label extension study.
- Part 3: Open-Label Extension 2: Following the successful completion of Part 2 of the study, eligible subjects could participate in Part 3, a 6-month open-label extension study.
- Overall: All treated subjects
Arm/Group | Part 1: Conversion | Part 2: Open-Label Extension 1 | Part 3: Open-Label Extension 2 | Overall
Serious Adverse Events (participants affected / at risk) | 1/43 | 5/32 | 3/12 | 9/43
Other Adverse Events (participants affected / at risk) | 18/43 | 17/32 | 9/12 | 35/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Conversion (N=43) | Part 2: Open-Label Extension 1 (N=32) | Part 3: Open-Label Extension 2 (N=12) | Overall (N=43)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Conversion (N=43) | Part 2: Open-Label Extension 1 (N=32) | Part 3: Open-Label Extension 2 (N=12) | Overall (N=43)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 0 (0) | 7 (7)
Upper Respiratory Infection (Infections and infestations) | 3 (3) | 5 (5) | 0 (0) | 8 (8)
Drug Toxicity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 2 (2) | 5 (5)
Dyskinesia (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 4 (4)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1) | 5 (5)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No